CLINICAL TRIAL: NCT01711281
Title: Monitoring of Hemodynamics in Heart Failure Patients by Intracardiac Impedance Measurement
Acronym: BIODetectHFII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR010
Record Dates: First submitted 2012-10-16; First posted 2012-10-22 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Implantable Cardioverter-Defibrillator; Intracardiac Impedance Measurement; Cardiac Resynchronization Therapy; Home Monitoring; Reverse Remodeling
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intracardiac Impedance Measurement (Experimental)
  Interventions: Device: Intracardiac Impedance Measurement Algorithm (integrated in CRT-D device)

INTERVENTIONS:
Device: Intracardiac Impedance Measurement Algorithm (integrated in CRT-D device)

SUMMARY:
Heart Failure (HF) is one of the most frequent diagnoses upon hospitalization and is a major cause of death. Cardiac resynchronization therapy (CRT) using an implantable device for synchronous bi-ventricular stimulation leads to improvement of hemodynamic parameters, physical capacity and quality of life. A continuous measurement of the left-ventricular volume would provide information about heart performance and could be used for both heart failure monitoring and optimization of CRT-therapy.

ELIGIBILITY:
Inclusion Criteria:

* De novo CRT-patients
* Planned implantation with a Lumax 740 HF-T device, a bipolar LV-lead and a true bipolar RV-lead
* NYHA class II or III
* QRS ≥ 150 ms
* LVEF between 15% and 35%
* LVEDD ≥ 55 mm
* Evaluable echo measurements

Exclusion Criteria:

* Persistent or permanent atrial fibrillation
* Heart surgery within the previous 3 months or planned for the time of study participation; post-heart transplantation or listed for heart transplantation
* Non-ambulatory patients
* Chronic renal dialysis
* Life expectancy less than 1 year due to a non-cardiac disease
* Age < 18 years and/or limited contractual capability
* Addiction to alcohol, medical drugs or illegal drugs
* Pregnant or breast-feeding women
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Intra-indivudual correlation coefficient r between stroke volume (SV) and stroke impedance (SZ). | Month 2
  SV will be assessed using Echo Doppler Ao-VTI (Aortic velocity time integral). SZ will be measured in parallel using intracardiac impedance measurement. The parameters will be assessed during a sequential measurement being conducted in month 2 of the observational period. Hemodynamic changes will be actively provoked using the CRT-D system for overdrive-pacing.

SECONDARY OUTCOMES:
Intra-individual correlation coefficient r between left-ventricular end-systolic volume (LVESV) and left-ventricular end-systolic impedance (LVESZ). | Month 2
  LVESV will be assessed using echo Biplane Simpson's method. LVESZ will be measured using the intracardiac impedance measurement. The parameters will be assessed during a sequential measurement being conducted in month 2 of the observational period. Hemodynamic changes will be actively provoked using the CRT-D system for overdrive-pacing.

OTHER OUTCOMES:
Intra-individual correlation coefficient r between stroke volume (SV) and stroke impedance (SZ). | Month 2
  SV will be assessed using a non-invasive blood pressure measurement device. SZ will be measured using the intracardiac impedance measurement.The parameters will be assessed during a sequential measurement being conducted in month 2 of the observational period. Hemodynamic changes will be actively provoked using the CRT-D system for overdrive-pacing.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sogaard, MD, PhD, Prof., Study Chair — Aalborg University, Aalborg University Hospital; Klaus-Jürgen Gutleben, MD, PhD, Study Chair — Herz- und Diabeteszentrum NRW, Bad Oeynhausen
Locations (22):
- Denmark (4):
  - Aalborg Sygehus, Kardiologisk Afdeling, Aalborg
  - Aarhus Universitetshospital, Hjertemedicinsk Afdeling B, Aarhus
  - Gentofte Hospital, Department P, Hellerup
  - Odense University Hospital, Hjertemedicinsk Afdeling B, Odense
- Germany (12):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charité Campus Virchow-Klinik, Medizinische Klinik mit Schwerpunkt Kardiologie, Berlin
  - Herzzentrum Brandenburg, Immanuel Klinikum, Bernau
  - Klinikum Bielefeld Mitte, Bielefeld
  - Evangelisches Krankenhaus, Bielefeld
  - Universitätsklinikum Essen, Westdeutsches Herzzentrum Essen, Essen
  - Medizinische Hochschule Hannover, Klinik für Kardiologie und Angiologie, Hanover
  - Kliniken Maria Hilf GmbH, Innere Medizin II, Klinik für Kardiologie, Mönchengladbach
  - Klinikum der Universität München - Grosshadern, München
  - Havellandklinik Nauen, Nauen
  - Krankenhaus Reinbek St. Adolf-Stift, Innere Abt. Kardiologie, Reinbek
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik I, Medizinische Intensiv- und Notfallmedizin, Würzburg
- Italy (2):
  - Azienda Ospedaliero Univesitaria, Ospedali Riuniti Umberto I- G.M. Lancisi- G. Salesi, Ancona
  - Fondazione Toscana G. Monasterio, Pisa
- Netherlands (3):
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - Isala Klinieken, Hospital de Weezenlanden, Department of Cardiology, Zwolle
- Universitätsspital Zürich, Zurich, Switzerland